CLINICAL TRIAL: NCT00074815
Title: Treatment of Pediatric OCD for SRI Partial Responders
Brief Title: Treatment of Obsessive Compulsive Disorder in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00008097; R01MH055121 (NIH); DSIR 84-CTM
Record Dates: First submitted 2003-12-19; First posted 2003-12-22 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2012-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Child; Adolescent
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Citalopram; Escitalopram; Fluoxetine; Fluvoxamine; Paroxetine; Clomipramine; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MedMgmt+CBT (Experimental): Participants will receive the following interventions: 1)SRI medication management with a psychiatrist plus, 2) cognitive behavioral therapy with a psychologist.
  Interventions: Drug: Serotonin reuptake inhibitors management; Behavioral: Cognitive behavioral therapy by a psychologist
- MedMgmt+I-CBT (Experimental): Participants will receive the following interventions 1)SRI medication management plus, 2) instructional cognitive behavioral therapy. Both of these will be implemented by the same psychiatrist.
  Interventions: Drug: Serotonin reuptake inhibitors management; Behavioral: Instructional cognitive behavioral therapy by a psychiatrist
- MedMgmt Only (Active Comparator): Participants will receive the intervention SRI medication management with a psychiatrist
  Interventions: Drug: Serotonin reuptake inhibitors management

INTERVENTIONS:
Drug: Serotonin reuptake inhibitors management — Participants are maintained on their optimized dose of SRI for OCD symptoms (see "Other Names" section for specific drugs and dosage ranges). If the participant has been treated with an SRI for at least 9 weeks AND has been at a stable dose for the past 3 weeks (e.g., the dose response curve is flat indicating no further improvement in OCD symptoms) OR the participant did not tolerate a dose increase to the next higher dose OR the participant has been at the maximum allowable dose for 3 weeks, then the participant is considered optimized and will be maintained on that dose. During trial, all participants will be maintained on their SRI dose during acute treatment at a constant dose unless side effects warrant downward adjustment of the SRI.
  Other Names: Drug Name with Minimum-Maximum Dosage; Citalopram (Celexa)10-60;; Escitalopram (Lexapro)5-30;; Fluoxetine (Prozac) 10-60;; Fluvoxamine (Luvox)25-300;; Paroxetine (Paxil)10-50;; Paroxetine-CR (Paxil)10-50;; Clomipramine (Anafranil)25-200;; Sertraline (Zoloft) 25-200;; Venlafaxine (Effexor)25-225;; Venlafaxine XR (Effexor)37.5-225;
Behavioral: Cognitive behavioral therapy by a psychologist — CBT consists of 14 visits over 12 weeks involving: (1) psychoeducation, (2), cognitive training, (3) mapping OCD, and (4) exposure and ritual prevention (EX/RP). The intervention was adapted from March and Mulle (1998) treatment protocol for pediatric OCD.
  Arms: MedMgmt+CBT
Behavioral: Instructional cognitive behavioral therapy by a psychiatrist — The psychiatrist who manages medication will also provide instructions in the CBT procedures that have been found to help reduce OCD symptoms, namely EX/RP. MM+I-CBT was constructed as a single-doctor "best practice" treatment with three primary goals: (1) inclusion of the main psychoeducational and EX/RP components of the full CBT protocol; (2) feasibility of training psychiatrists to perform the CBT component of MM+I-CBT; (3) integration with protocol medication management visits; and (4) feasibility of implementation with the constraints of a busy practice oriented primarily toward pharmacotherapy.
  Arms: MedMgmt+I-CBT

SUMMARY:
This study will determine whether cognitive behavioral therapy delivered by either psychologists or psychiatrists can improve the effectiveness of serotonin reuptake inhibitor treatment in children with obsessive compulsive disorder.

DETAILED DESCRIPTION:
The vast majority of children with obsessive compulsive disorder (OCD) are given serotonin reuptake inhibitor (SRI) drugs as initial treatment. However, recommended doses of these medications leave many children with clinically significant residual symptoms. Health care experts typically recommend augmenting SRI treatment with cognitive behavioral therapy (CBT), yet this recommendation is seldom followed. This study will contrast two CBT augmentation strategies to continued medication management alone: CBT administered by a psychologist and instructional CBT (I-CBT)administered by a psychiatrist in the context of ongoing medication management.

All patients in the trial will be eligible to receive a full course of CBT by study end. Participants in this study will be randomly assigned to receive CBT, I-CBT or continued medication management. All participants will continue their SRI treatment for 12 weeks. After the 12-week treatment period, participants who received I-CBT or medication management alone and who remain symptomatic will be given CBT as will participants who are asymptomatic but relapse within 6 months after treatment. Assessments will be conducted at Weeks 0, 4, 8, and 12. Follow-up assessments will be conducted at 3 and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Diagnosis of obsessive compulsive disorder
* CYBOCS total score greater than 16

Exclusion Criteria:

* Other primary or co-primary psychiatric disorder
* Pervasive developmental disorder or disorders, including Asperger's Syndrome
* Thought disorder
* Prior failed trial of cognitive-behavioral therapy
* Has pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS) or maintenance antibiotic for obsessive-compulsive disorder
* Mental retardation
* Pregnancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2003-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S March, MD MPH, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Child and Family Study Center, Durham, North Carolina
  - University of Pennsylvania, The Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Franklin ME, Sapyta J, Freeman JB, Khanna M, Compton S, Almirall D, Moore P, Choate-Summers M, Garcia A, Edson AL, Foa EB, March JS. Cognitive behavior therapy augmentation of pharmacotherapy in pediatric obsessive-compulsive disorder: the Pediatric OCD Treatment Study II (POTS II) randomized controlled trial. JAMA. 2011 Sep 21;306(11):1224-32. doi: 10.1001/jama.2011.1344. PMID 21934055
- [Derived] Conelea CA, Selles RR, Benito KG, Walther MM, Machan JT, Garcia AM, Sapyta J, Morris S, Franklin M, Freeman JB. Secondary outcomes from the pediatric obsessive compulsive disorder treatment study II. J Psychiatr Res. 2017 Sep;92:94-100. doi: 10.1016/j.jpsychires.2017.04.001. Epub 2017 Apr 7. PMID 28412602
- [Derived] Conelea CA, Walther MR, Freeman JB, Garcia AM, Sapyta J, Khanna M, Franklin M. Tic-related obsessive-compulsive disorder (OCD): phenomenology and treatment outcome in the Pediatric OCD Treatment Study II. J Am Acad Child Adolesc Psychiatry. 2014 Dec;53(12):1308-16. doi: 10.1016/j.jaac.2014.09.014. Epub 2014 Oct 2. PMID 25457929
- [Derived] Freeman JB, Choate-Summers ML, Garcia AM, Moore PS, Sapyta JJ, Khanna MS, March JS, Foa EB, Franklin ME. The Pediatric Obsessive-Compulsive Disorder Treatment Study II: rationale, design and methods. Child Adolesc Psychiatry Ment Health. 2009 Jan 30;3(1):4. doi: 10.1186/1753-2000-3-4. PMID 19183470

RESULTS

PARTICIPANT FLOW:
Groups:
- MM + CBT: Participants will receive medication management plus cognitive behavioral therapy with a psychologist
- MM + ICBT: Participants will receive medication management plus instructional cognitive behavioral therapy with a psychiatrist
- MM Only: Participants will receive medication management only
Period: Overall Study
Arm/Group | MM + CBT | MM + ICBT | MM Only
Started | 42 | 40 | 42
Completed | 37 | 34 | 30
Not Completed | 5 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MM + CBT | MM + ICBT | MM Only | Total
Number analyzed (Participants) | 42 | 40 | 42 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 40 | 42 | 124
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.71 (2.88) | 13.76 (2.72) | 14.34 (2.51) | 13.6 (2.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 22 | 66
  Male | 19 | 19 | 20 | 58
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 42 | 124

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: OCD symptom severity was measured using the CY-BOCS, an interviewer-rated instrument that assess obsessions and compulsions separately on time consumed, distress, interference, degree of resistance, and control; it yields separate severity scores for obsessions and for compulsions (0 - 20), and a composite symptom severity score (0 to 40).
  Consistent with signal detection analyses examining the optimal criterion for treatment response, a CY-BOCS reduction of 30% or more from baseline to week 12 was used as the criterion for RESPONSE and was the primary dichotomous outcome measure.
Time Frame: Measured at baseline and Week 12.
Population: Intent to treat (all included)
Measure: Number (95% Confidence Interval); unit: Proportion of Participants with RESPONSE
Arm/Group | MM + CBT | MM + ICBT | MM Only
Number analyzed (Participants) | 42 | 40 | 42
Proportion of Participants with RESPONSE | 0.69 [0.54 to 0.83] | 0.34 [0.18 to 0.50] | 0.30 [0.15 to 0.45]

2. Secondary Outcome: Child Obsessive -Compulsive Impact Scale (COIS)
Time Frame: Measured at baseline; Weeks 4, 8, and 12; and Months 3 and 6 of follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Child Depression Inventory
Time Frame: Measured at baseline; Weeks 4, 8, and 12; and Months 3 and 6 of follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Pediatric Adverse Event Rating Scale (PAERS)
Time Frame: Measured at baseline; Weeks 4, 8, and 12; and Months 3 and 6 of follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | MM + CBT | MM + ICBT | MM Only
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/40 | 1/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MM + CBT (N=42) | MM + ICBT (N=40) | MM Only (N=42)
Suicide Attempt that led to hospitalization and changes to medication and therapy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Attempt led to premature termination of treatment protocol (i.e., additional treatment outside of randomized treatment protocol). Stopped OCD treatment and began treating subject's comorbid depression.
Suicidal Thoughts due to school difficulties (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — In last protocol session, subject reported suicidal thoughts due to teasing by classmates. Given the context in which these thoughts arose (social difficulties at school), this serious adverse event was determined to be unrelated to treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No